CLINICAL TRIAL: NCT04117295
Title: Carmat Total Artificial Heart Early Feasibility Study
Brief Title: Carmat TAH Early Feasibility Study
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Occurrence of a quality issue affecting some of its prostheses
Sponsor: Carmat SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR2019-US
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: End-stage Heart Failure
Keywords: Heart Replacement Therapy; Total Artificial Heart; Biventricular Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Subjects implanted with the Carmat TAH
  Interventions: Device: Carmat Total Artificial Heart

INTERVENTIONS:
Device: Carmat Total Artificial Heart — Heart replacement therapy

SUMMARY:
Feasibility study of the Carmat TAH as a treatment for transplant-eligible patients in severe, end-stage heart failure.

DETAILED DESCRIPTION:
This is a prospective, multi-center, staged feasibility study designed to assess the initial evidence of safety and performance of the Carmat TAH in the treatment of severe, end-stage heart failure. This study will include up to 7 centers in the US. The study population will include up to 10 transplant-eligible patients enrolled and implanted with the Carmat TAH.

Data collection will be recorded prior to implantation of the device and for six months following implant, then long term at 9, 12, 18 and 24 months while the patient remains on the device. Adverse events, as defined by INTERMACS, while on device support will be collected throughout the study until study closure and will be adjudicated by an independent Clinical Event Committee.

Progress reports of the clinical outcomes will be reviewed by the DSMB after implantation of each patient and every three months thereafter while any patient is supported with the device. A progress report will be sent to FDA for review after three subjects have been implanted and followed for 60 days.

The primary objective of the study is survival on an original Carmat device at 180 days post-implant or survival to cardiac transplantation if occurring before 180 days post-implant.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years of age or older at the time of informed consent
2. Anatomic compatibility confirmed using 3D imaging (CT-scan).
3. Inotrope dependent (with documented attempt to wean) or cardiac Index (CI) < 2.2 L/min/m2 if inotropes are contra-indicated (heart failure due to restrictive or constrictive physiology).
4. On Optimal Medical Management as judged by the investigator based on current Heart Failure practice guidelines (ESC/AHA).
5. Eligible for biventricular Mechanical Circulatory Support according to ISHLT guidelines for mechanical circulatory support:

   1. Biventricular failure with at least two of the following hemodynamic/ echocardiographic measurements implying right heart failure: RVEF ≤30%; RVSWI ≤0.25mmHg*L/m2; TAPSE ≤14mm; RV-to-LV end-diastolic diameter ratio >0.72; CVP >15 mmHg; CVP-to-PCWP ratio >0.63; Tricuspid insufficiency grade 4; PAPi<2
   2. Treatment-refractory recurrent and sustained ventricular tachycardia or ventricular fibrillation in the presence of untreatable arrhythmogenic pathologic substrate.
   3. Heart failure due to restrictive or constrictive physiology (e.g., hypertrophic cardiomyopathy, cardiac amyloidosis / senile or other infiltrative heart disease).
6. Patient has signed the informed consent, has full understanding of procedures, and is committed to following study requirements.
7. Eligible for cardiac transplantation

Exclusion Criteria:

1. Known intolerance to anticoagulant or antiplatelet therapies or known Heparin Induced Thrombocytopenia.
2. Presence of any non-temporary mechanical circulatory support
3. Presence of temporary mechanical circulatory support such as Impella (all types) or IABP with a duration greater than 21 days
4. Presence of ECMO with a duration greater than 7 days
5. Patient is intubated and unconscious, or intubated and not awake
6. Coagulopathy defined by platelets < 100k/µl or INR ≥ 1.5 not due to anticoagulant therapy.
7. Cerebrovascular accident < 3 months or symptomatic or a known > 80% carotid stenosis.
8. Known abdominal or thoracic aortic aneurysm > 5 cm that has not been treated.
9. Severe end-organ dysfunction as per any of the following criteria:

   1. Total bilirubin > 2.5 mg/dl or cirrhosis evidenced by ultrasound, CT-scan and positive biopsy
   2. eGFR < 30ml/min/1.73m2 or the need for chronic renal replacement therapy
10. History of severe Chronic Obstructive Pulmonary Disease with FEV1/FVC <0.7, or FEV1<50% predicted or severe restrictive lung disease.
11. Recent blood stream infection (<7 days).
12. Documented amyloid light-chain (AL amyloidosis).
13. Hemodynamically significant peripheral vascular disease with documented ankle- brachial pressure index (ABPI) <0.3.
14. Illness, other than heart disease, that would limit survival to less than 2 years.
15. Irreversible cognitive dysfunction, psychosocial issues or psychiatric disease, likely to impair compliance with the study protocol and TAH management that in the opinion of the investigator could interfere with the ability to manage the therapy (i.e. non-compliance to heart failure therapy, uncontrolled diabetes, mental health issue, etc.).
16. Current or planned pregnancy or breast feeding (woman of childbearing age will have to show negative pregnancy test).
17. Patient is currently enrolled or has participated in the last 30 days in another therapeutic or interventional clinical study that is likely to confound the study results or affect the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 180 days
  Proportion of patients surviving on the Carmat TAH

SECONDARY OUTCOMES:
Survival without Permanent Neurologic Deficit | 180 days
  Proportion of patients surviving post implant without a permanent disabling stroke (Modified Rankin Scale >3)
Post transplant survival | 30 days
  Proportion of patients surviving 30 days post-transplant
Change in functional status | 180 days
  New York Heart Association (NYHA) functional classification (regression scale I, II, III, IV)
Change in functional status measured by the Six Minutes Walk Test | 180 days
  The 6-min walk test is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Generic health status change | 180 days
  Measured with the EuroQol EQ-5D questionnaire, a descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses (EQ-5D-5L). The responses record five levels of severity (1:no problems; 2:slight problems; 3:moderate problems 4:severe problems; 5:extreme problems) within a particular EQ-5D dimension.
  Measured with the Kansas City Cardiomyopathy Questionnaire, a self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Adverse Events | 180 days
  Adverse Event Rates will be captured per the INTERMACS definitions
Hospital readmission rate | 180 days
  Rate of unplanned readmissions to the hospital

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Louisville Jewish Hospital, Louisville, Kentucky
  - Duke University Medical Center, Durham, North Carolina
  - Baylor University Medical Center, Dallas, Texas
  - VCU Medical Center, Richmond, Virginia